CLINICAL TRIAL: NCT02582853
Title: sCD163 as a Potential Biomarker in Guillain- Barré Syndrome
Acronym: GBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: GBS CD163; 1-10-72-256-15 (Other: The National Committee on Health Research Ethics (Denmark)); 1-16-02-522-15 (Other: The Danish Data Protection Agency)
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Guillain-Barre Syndrome
Keywords: GBS; AIDP; Spinal fluid; sCD163
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Spinal Puncture; Blood Specimen Collection

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Spinal fluid and blood sample for identification of different factors
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients diagnosed with GBS: Patients will undergo a lumbar puncture as a part of the diagnostic procedure as soon as they are suspected to be suffering from GBS on clinical grounds with blood test. The procedure and a blood test will be repeated after 6 months.
  Lumbar puncture Blood sample
  Interventions: Procedure: Lumbar puncture; Procedure: Blood Sample
- Symptomatic controls: Controls include patients with unspecified neurological symptoms or diseases who will undergo a lumbar puncture at the Department of Neurology at Aarhus University Hospital as part of their diagnostic work up irrespective of this study. We expect to include 40 symptomatic controls.
  Interventions: Procedure: Lumbar puncture; Procedure: Blood Sample

INTERVENTIONS:
Procedure: Lumbar puncture — Lumbar puncture for spinal fluid
  Other Names: Spinal tap
Procedure: Blood Sample — Blood sample

SUMMARY:
Guillain- Barré syndrome (GBS) is an acute inflammatory demyelinating polyneuropathy (AIDP) that often is triggered by an infection. GBS is characterized by progressing weakness and numbness and loss of tendon of reflexes. It can also include tingling sensation in the legs and arms. These symptoms occur due to an autoimmune attack on the myelin resulting in demyelination.

The diagnosis is given by electrophysiological examination and clinical presentation.

GBS is treated with intravenous immunoglobulin (IVIG) and plasma exchange (PE). Both treatments are equally effective. Most patients recover completely, while others must ease symptoms and reduce the duration of illness by several treatments.

The purpose of this study is to define if patients with GBS have higher concentrations of sCD163 in their cerebrospinal fluid and serum compared with symptomatic control subjects. Furthermore it is to define if the concentrations of sCD163 reduces after treatment.

DETAILED DESCRIPTION:
Guillain- Barré syndrome (GBS) is an acute inflammatory demyelinating polyneuropathy (AIDP) that often is triggered by an infection. GBS is characterized by progressing weakness and numbness and loss of tendon reflexes. It can also include tingling sensation in the legs and arms. These symptoms occur due to an autoimmune attack on the myelin resulting in demyelination. The diagnosis is given by electrophysiological examination and clinical presentation. GBS is treated with intravenous immunoglobulin (IVIG) or plasma exchange (PE). The specific mechanism is not fully understood, but it is believed that the antibodies produced against the myelin, is eliminated to avoid further damage to the peripheral nerves. IVIG is slightly safer and easier to give than PE. However, both treatments are equally effective. They both need to be given during the first few weeks of symptoms.

Most patients recover completely, while others must ease symptoms and reduce the duration of illness by several treatments. Moreover, the initial phase of GBS is followed by a long recovery period where intensive neurorehabilitation is important. Some people will not recover completely from GBS and experience long-term complications such as not being able to walk unaided, loss of sensation causing lack of coordination and balance. It is estimated around 20% of people with GBS still experience some muscle weakness after three years. Some may also have persistent fatigue. In rare cases, complications can be life threatening, particularly in the acute phase.

GBS is one of the neurological emergencies, where patients need to be examined closely during the initial acute phase of the illness. Many studies have been performed to elucidate the mechanism of neuropathy in Guillain Barré syndrome but treatment remains disappointing. There are findings of autoantibodies against gangliosides, myelin proteins such as PO- glycoprotein, P2 basic protein and PMP22 and to nodal and paranodal proteins, such as NF155 and NF186.

Cluster of differentiation 163 (CD-163) - a new way to measure GBS CD-163 is a scavenger receptor (recognizes and uptakes macromolecules), which marks the monocyte-macrophage activation. CD163 works for macrophages as a receptor for haemoglobin-haptoglobin complexes. The soluble form of the receptor is called sCD163 and is found in plasma, where it is up regulated in a large range of inflammatory diseases.

Values, which are increased strongly (<20mg/l), are seen in diseases like macrophage activating syndrome, haemophagocytic syndrome and acute hepatic failure. Furthermore, the level of sCD163 reflects the activity of the disease. Patients with increasing and high values are found to have unfavourable prognosis. Increased values (5-20 mg/l) are seen in hepatic disease, sepsis and Gaucher´s disease. Septic patients with values greater than 10mg/l have a 10 times greater risk of fatal outcome. Values, which are slightly increased (3-5 mg/l), are often seen in inflammatory of infectious conditions and in cancer.

Purpose and Hypothesis Purpose To define the concentration of sCD163 in the cerebrospinal fluid and serum in patients with GBS patients compared with controls.

The project hypothesis Our hypothesis is that the inflammatory biomarker sCD163 is increased in CSF and blood from GBS patients compared to controls Perspectives Due to the various clinical variants of inflammatory polyneuropathies and due to the lack of biomarkers, it remains difficult to diagnose GBS. It is very important to identify new methods for diagnosis and monitoring of patients with GBS. This may also enable better prediction of the prognosis and the level of treatment needed.

The pathology of GBS is still unknown but it is known to be immune mediated. In several studies sCD163 has been shown to up regulated in a larger range of inflammatory diseases suggesting sCD163 to be a relevant biomarker for GBS.

Study population

The study population will consist of two subgroups:

1. Patients diagnosed with GBS Patients will undergo a lumbar puncture as a part of the diagnostic procedure as soon as they are suspected to be suffering from GBS on clinical grounds with blood test. The procedure and a blood test will be repeated after 6 months.
2. Symptomatic controls Controls include patients with unspecified neurological symptoms or diseases who will undergo a lumbar puncture at the Department of Neurology at Aarhus University Hospital as part of their diagnostic work up irrespective of this study. The investigators expect to include 40 symptomatic controls.

Due to admission to the Department of Neurology, Aarhus University Hospital with the diagnosis of suspected GBS all eligible participants will receive information about the project and will be asked to give their consent to participation.

As mentioned the controls are recruited patients, who nevertheless will undergo lumbar puncture for another reason to the Department of Neurology, will be informed about the project and will be asked to participate. Control patients will be participating only once.

The investigators anticipate including 20 patients with GBS and 40 symptomatic controls.

Participants will receive written and oral information about the study. The oral information will take place at Department of Neurology, Aarhus University Hospital. Moreover, the pamphlet " Før du deltager i et sundhedsvidenskabeligt forsøg"(about participating in a clinical trial) will be handed out.

The information will be given by consultant Henning Andersen, MD Lars Markvardsen or stud. med. Malalai Musleh. It is possible for the participants to bring a companion and they are offered about an hour to consider the participation because the procedure of lumbar puncture will take place at the same day. If the patient need to consider the participation with a companion and it is not possible for the participants to bring a companion within an hour, then they will not be included in the study.

The participants will be informed of that information from the medical record will be passed on and included and used in this project including past medical history, actual use of drugs, results of biochemical analyses and brain imaging, abnormalities at the clinical examinations and the conclusions from the doctors diagnostic workup.

If new knowledge about disadvantages of participating in the study appears the participants will be informed immediately.

Moreover, the participant will be informed if evaluations during the study bring knowledge about the general health status of the patient, unless this has been clearly rejected by the patient.

By the end of the study it is possible for participants to contact the study coordinator to get information about study results.

Method All source data from the study will be stored according to Danish legislation and the study will be approved by the Danish Data Protection Agency.

Lumbar puncture and Serum The participation implies extraction 2-3 ml of spinal fluid and a blood sample about 10 ml, which will be used for analysis of sCD163. Spinal fluid and blood samples will be drawn in the same procedure as the diagnostic samples. For the GBS patients a repeat blood test will be performed after 2-4 weeks and again after 6 months. The extraction of blood sample will be about 10 ml each repeated test. A repeated lumbar puncture will be performed after 6 months as well, where the extraction amount will also be about 2-3ml of spinal fluid. The patients have full right to say no to the repeated procedure. The symptomatic controls will only have spinal fluid and blood samples drawn once.

Other examinations

Patients with GBS will undergo a clinical examination with the following the neuropathy scores:

Participants will be evaluated clinically with: Neuropathy Impairment Score (NIS):

The NIS is a composite clinical scoring system that has been widely used to objectively assess the severity of peripheral neuropathy. The NIS quantifies the findings of the neurologic examination by attributing a score (ranging from 0 [normal] to 88 [total impairment]) to the clinical abnormalities noted in the physical assessment of sensation, muscle power, and tendon reflexes.

Overall Disability Sum Score (ODSS):

The ODSS seems to be valid and sensible measure to score dysfunction and disability in patients with motor neuropathies. This score is composed of arm and leg disability scale with a total score ranging from 0 (no signs of disability) to 12 (most severe disability score). The patient and the observer will judge each activity with: not affected, affected and not prevented or prevented.

Analyses The spinal fluid and the serum will be analysed at the Medical Research Laboratory. The spinal fluid and blood samples will be deposited in a research biobank at Aarhus University Hospital. The plan is to carry out all the biochemical analyses at the same time when all samples are collected. Any excess biological material will be transferred to a biobank for future research.

Serum and CSF will be analyzed for sCD163 and other inflammatory markers, by already established techniques at the Department of Clinical Medicine, Aarhus University Hospital and the spinal fluid will be examined with spectrometry.

Statistics GBS is a rare disease and because of the low number of patients, it is difficult to perform power calculations in studies of GBS patients. However, the investigators anticipate that 20 patients and 40 controls will be sufficient.

The program STATA will be used for statistical analyses. Parametric or non- parametric tests will be used depending of the normal distribution of data. In all statistical analysis a 5% level of significance will be used.

Ethical considerations The local Ethics Committee of the Central Region of Denmark will approve the study.

The tests performed on the patients involved in this research project are lumbar puncture, blood sampling and clinical examination.

A lumbar puncture is a procedure used to collect cerebral spinal fluid (CSF) for analysis. CSF is a promising source of biomarkers in GBS since the proximal nerve roots, which are affected early in the disease, are in close anatomical contact with the CSF space.

During the procedure a hollow needle is used to penetrate the spinal canal at the level of the third- to-fourth or fourth-to-fifth lumbar vertebra in the low back. CSF then drips out through the needle and is collected. It involves some risk to perform a lumbar puncture, which include post lumbar puncture headache with an incidence of 12%, most common in younger patients. Most frequently, the headache has a short duration and it may be cured with application of a blood -patch. Moreover, lumbar puncture can cause temporary lumbar pain and an accumulation of blood underneath the skin. There is a very low risk of bleeding in the epidural space with compression of spinal nerves and an even lower risk of infections (meningitis or meningoencephalitis).

However, it is important to highlight that lumbar puncture will be performed as a routine diagnostic for GBS patients; therefore it will not cause the participants any further problem.

The investigators consider this project to be ethically acceptable considering of the low risk involved in this project, the seriousness and costs of the disease and the potential to identify a relevant biomarker in GBS.

At all times during the diagnostic work-up and consequently in the research project investigators will do this with respect for the patients mental and physical condition. The research project will be carried out according to the Act on Processing of Personal Data and, furthermore, the project will be submitted to the common regional information system for Region Midtjylland Publications Positive, negative or inconclusive results will be published in an international journal with Malalai Musleh as first author, Professor Henning Andersen as senior author and Lars Markvardsen will be co-author.

ELIGIBILITY:
Inclusion Criteria:

* Progressive muscle weakness with acute onset (< 2 weeks)
* Areflexia

Exclusion Criteria:

* Other cause of peripheral neuropathy
* Malignant disease
* Age < 18 years
* Unable to give informed consent
* Ongoing infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of two groups:
  1. Patients diagnosed with GBS
  2. Symptomatic controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of sCD163 in patients with GBS | Day 1

SECONDARY OUTCOMES:
Concentration of sCD163 in patients with GBS after treatment | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, Professor, Principal Investigator — Department of Neurology
Locations (1):
- The Department of Neurology, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Background] Haunsø, Stig m.fl.: Medicinsk Kompendium: 18. Udgave, Nyt Nordisk forlag, 2013
- [Background] Bourque PR, Chardon JW, Massie R. Autoimmune peripheral neuropathies. Clin Chim Acta. 2015 Sep 20;449:37-42. doi: 10.1016/j.cca.2015.02.039. Epub 2015 Mar 4. PMID 25748038
- [Background] Fuglsang-Frederiksen A, Pugdahl K. Current status on electrodiagnostic standards and guidelines in neuromuscular disorders. Clin Neurophysiol. 2011 Mar;122(3):440-455. doi: 10.1016/j.clinph.2010.06.025. Epub 2010 Jul 31. PMID 20673740
- [Background] Moller HJ. Soluble CD163. Scand J Clin Lab Invest. 2012 Feb;72(1):1-13. doi: 10.3109/00365513.2011.626868. Epub 2011 Nov 7. PMID 22060747
- [Background] Etzerodt A, Moestrup SK. CD163 and inflammation: biological, diagnostic, and therapeutic aspects. Antioxid Redox Signal. 2013 Jun 10;18(17):2352-63. doi: 10.1089/ars.2012.4834. Epub 2012 Oct 19. PMID 22900885
- [Background] Kjaergaard AG, Rodgaard-Hansen S, Dige A, Krog J, Moller HJ, Tonnesen E. Monocyte expression and soluble levels of the haemoglobin receptor (CD163/sCD163) and the mannose receptor (MR/sMR) in septic and critically ill non-septic ICU patients. PLoS One. 2014 Mar 17;9(3):e92331. doi: 10.1371/journal.pone.0092331. eCollection 2014. PMID 24637679
- [Background] Merkies IS, Schmitz PI, van der Meche FG, Samijn JP, van Doorn PA; Inflammatory Neuropathy Cause and Treatment (INCAT) group. Clinimetric evaluation of a new overall disability scale in immune mediated polyneuropathies. J Neurol Neurosurg Psychiatry. 2002 May;72(5):596-601. doi: 10.1136/jnnp.72.5.596. PMID 11971045